CLINICAL TRIAL: NCT00422279
Title: Evaluation of Implant Stability and Local Bone Formation at Endosseous Dental Implants With a Titanium Porous Oxide Surface Adsorbed With rhBMP-2
Brief Title: A Study of Dental Implants Coated With Bone Morphogenetic Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR06:3393
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Alveolar Ridge Abnormality
Keywords: Bone Inductive Implant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supraalevolar (Experimental): Bone inductive implant (Nobel Replace Tapered Groovy) placed in the supralveolar position
  Interventions: Device: Nobel Replace Tapered Groovy
- Other (Experimental): Bone inductive implant (Nobel Replace Tapered Groovy) placed in extraction socket
  Interventions: Device: Nobel Replace Tapered Groovy

INTERVENTIONS:
Device: Nobel Replace Tapered Groovy — Bone inductive implant placed in supralveoral position or extraction site
  Other Names: Bone inductive implant

SUMMARY:
The purpose of the study is to evaluate implant stability and stimulate clinically relevant horizontal and vertical new bone formation around Nobel Biocare's Bone Inductive Implant.

DETAILED DESCRIPTION:
Common complications encountered when replacing missing teeth with Endosseous dental implants include lack of adequate bone volume limiting the possibility of optimal patient treatment. Typical limitations include severely resorbed alveolar ridges (height and width) in patients following long-term edentulism. In other cases, the alveolar ridge may have become compromised due to advanced periodontal disease, traumatic extractions, and other trauma disallowing Endosseous dental implant placement to meet aesthetic and functional demands. Conversely, placing Endosseous dental implants to optimally meet aesthetic and functional demands in sites exhibiting alveolar ridge aberrations often results in partial exposure of the Endosseous dental implant bone-anchoring surface. In some cases clinicians have attempted to overcome the deficient bone volume by augmenting the anticipated Endosseous dental implant site using bone biomaterials, commonly originating from human or animal cadaveric sources, or synthetic biomaterials. The biomaterials have been used alone and in combinations including autologous bone grafts. Non-resorbable and bioresorbable barrier devices have been used to prevent dislocation of implanted biomaterials. The ability of the Bone Inductive Implant to form new bone above the level of the resorbed alveolar ridge to immerse the exposed portion of the Endosseous dental implant in bone (Treatment group 1) and the ability of the Bone Inductive Implant to induce bone formation around stable Endosseous dental implants placed into tooth extraction sockets (Treatment group 2) without the use of bone grafts, bone biomaterials, or barrier devices will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18 years.
* 2 teeth or more are missing either upper/lower jaw (Treatment Gp 1)
* 2 or more teeth require extraction either upper/lower jaw.(Treatment Gp 2)

Exclusion Criteria:

* Medical risk patients
* Smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PHILIP J HANES, DDS, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Becker W, Wikesjo UM, Sennerby L, Qahash M, Hujoel P, Goldstein M, Turkyilmaz I. Histologic evaluation of implants following flapless and flapped surgery: a study in canines. J Periodontol. 2006 Oct;77(10):1717-22. doi: 10.1902/jop.2006.060090. PMID 17032115
- [Result] Wikesjo UM, Susin C, Qahash M, Polimeni G, Leknes KN, Shanaman RH, Prasad HS, Rohrer MD, Hall J. The critical-size supraalveolar peri-implant defect model: characteristics and use. J Clin Periodontol. 2006 Nov;33(11):846-54. doi: 10.1111/j.1600-051X.2006.00985.x. Epub 2006 Sep 11. PMID 16965525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four patients have been recruited to participate in this study after they met the inclusion criteria, all patients have been recruited at the Medical college of Georgia, Augusta, GA, USA
Pre-assignment Details: all the four study patients met the inclusion criteria no run in's have been encountered, all the patients completed this study at the scheduled follow up visits
Groups:
- Supraalveolar Position: bone inductive implants (Nobel Replace Tapered Groovy) placed in supraalveolar position
- Extraction Sites: bone inductive implants (Nobel Replace Tapered Groovy) placed in tooth extraction sockets
Period: Overall Study
Arm/Group | Supraalveolar Position | Extraction Sites
Started | 2 | 2
24 Month After Loading Period | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Supralveolar Position: bone inductive implants placed in supraalveolar position
- Extraction Sites: bone inductive implants placed in tooth extraction sites
- Total: Total of all reporting groups
Arm/Group | Supralveolar Position | Extraction Sites | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Showing Bone Growth With rhBMP-2 (15 and 30 µg Per Implant)
Description: The secondary endpoint of the study was to assess the minimum dose of rhBMP2 eliciting bone growth.The secondary endpoint was assessed by measuring using a probe the quantity of any newly formed bone 1.in the group where implants were placed in the supra alveolar position the treatment is successful if the bone exceeds 1.5 mm above the initial alveolar bone level in all measured points 1. in the group where implants were placed in extraction sockets the treatment is successful if the gap between the implant body and the extraction socket is filled with Bone.
  Safety dose used:- In the dog model; seroma formation was extensive with higher rhBMP-2 concentrations (3.0 and 4.0 mg/mL.Seromas was also significant in the dog model for the 0.75 and 1.5 mg/mL rhBMP-2 concentrations, hence a minimum dose of 15 and 30 µg per implants was chosen)
Time Frame: 3 months
Population: 1.When implants were placed in the supraalveolar position the treatment was not successful 2. in the group where implants were placed in extraction sockets the treatment was not successful
Measure: Number; unit: Number of participants with bone grow
Groups:
- Supra Aleveolar Position: bone inductive implants (Nobel Replace Tapered Groovy) placed in supraalveolar position
Arm/Group | Supra Aleveolar Position | Extraction Sites
Number analyzed (Participants) | 2 | 2
Number of participants with bone grow | 0 | 0

2. Primary Outcome: Primary Endpoint Was to Assess Implant Stability of the Implants( 4 Patients in Two Groups With a Total of 8 Implants) at Baseline and After 3 Months of Submerged Healing and After 6 Months of Prosthetic Loading
Description: The following success criteria for the primary endpoint have been adopted and apply to both treatment groups. 1.The implant stability (ISQ) was recorded by means of resonance frequency analysis (RFA) at implant insertion, 3 months and after 6 months of loading 2. radiographic and computed tomography analyses shall not show any signs of peri-implant radiolucency at the 3 and 6 month time point 3. implant stability after 3 months shall allow tightening to 35Ncm without implant rotation by using a torque wrench
Time Frame: Implant insertion, 3 months, 6 months
Population: Implant stability was measured using a torque wrench, Resonance frequency analysis was conducted, radiographs were analyzed and computed tomography was performed
Measure: Number; unit: implants
Units Other Than Participants: Implants
Groups:
- Supraalveloar Postion: bone inductive implants placed in supraalveolar position a total of 2 patients with 4 implants ( two implants in each patient)
- Extraction Sites: bone inductive implants placed in tooth extraction sockets with a total of 2 patients with 4 implants ( two implants in each patient)
Arm/Group | Supraalveloar Postion | Extraction Sites
Number analyzed (Participants) | 2 | 2
Number analyzed (Implants) | 4 | 4
implants
  Stability Baseline | 4 | 4
  Stability 3 months submerged healing | 4 | 3
  Stability 6 months Prosthetic loading | 4 | 3

ADVERSE EVENTS:
Groups:
- Supralveolar Position: bone inductive implants (Nobel Replace Tapered Groovy) placed in supraalveolar position
- Extraction Sites: bone inductive implants (Nobel Replace Tapered Groovy) placed in tooth extraction sites
Arm/Group | Supralveolar Position | Extraction Sites
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supralveolar Position (N=2) | Extraction Sites (N=2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) — Subject 03 was diagnosed with hyperthyroidism 2 weeks prior to the visit and had started medication (Tapazole and Inderol).
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject 04 reported that she had been diagnosed to suffer from osteoporosis prior to the study. During the first 1½ to 2 months of implant treatment she did not receive medication but later began bisphosphonate drugs (Boniva, 200 mg, po, monthly);

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
I understand that I retain the right to publish the data from the clinical work that I perform. I agree that Nobel Biocare USA, LLC will be allowed to review and comment on such a document prior to its publication to ensure that the document does not disclose any trade secrets or other confidential information which may be known to me by virtue of my participation in the clinical study. I will not disclose any information regarding the study without permission from Nobel Biocare USA, LLC.